CLINICAL TRIAL: NCT06014658
Title: A Multicenter, Open-label, Phase 1/1b / Phase 2 Dose Finding, Safety, and Pharmacokinetic Study of MBRC-101, an Anti-EphA5 Monomethyl Auristatin E (MMAE) Antibody Drug Conjugate, in Advanced Refractory Solid Tumors
Brief Title: Safety, PK, and Preliminary Efficacy of MBRC-101 in Advanced Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MBrace Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MBRC-101-001
Record Dates: First submitted 2023-08-01; First posted 2023-08-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Immunoconjugates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Dose Escalation (Experimental)
  Interventions: Drug: Antibody-Drug Conjugate
- Phase 1b Expansion (Experimental)
  Interventions: Drug: Antibody-Drug Conjugate
- Phase 2 (Experimental)
  Interventions: Drug: Antibody-Drug Conjugate

INTERVENTIONS:
Drug: Antibody-Drug Conjugate — MBRC-101: AN ANTI-EPHA5 MONOMETHYL AURISTATIN E (MMAE) ANTIBODY DRUG CONJUGATE

SUMMARY:
This is a first-in-human (FIH), open label Phase 1/1b / Phase 2 study in patients with advanced metastatic solid tumors refractory to standard treatment. Phase 1 will identify potential optimal biologically relevant doses (OBRD) and the maximum tolerated dose (MTD) of MBRC-101 at one 1 or more dosing regimens. Phase 1b will evaluate the safety and preliminary clinical activity of MBRC-101 at potential OBRDs. Phase 1 and Phase 1b will both characterize single and multiple-dose PK profiles and evaluate incidence and persistence of anti-MBRC-101 Ab. Phase 2 will evaluate the efficacy of MBRC-101 at the RP2D from Phase1b.

DETAILED DESCRIPTION:
Phase 1, dose escalation, will enroll approximately 30 patients with advanced or metastatic solid tumors refractory to standard therapy. EphA5 expression will not be required for enrollment into Phase 1 but will be assessed retrospectively.

Phase1b, the dose expansion phase will evaluate the safety and preliminary clinical activity of MBRC-101 at potential OBRDs and dosing regimens in patients with advanced or metastatic solid tumors refractory to standard therapy. Phase 1b will enroll 3 expansion cohorts of ≈ 20 patients per cohort (n ≈ 60 total).

The Phase 2 portion will begin when the RP2D has been determined from Phase 1b and all Phase 1b patients have completed at least two cycles of treatment or have discontinued from the study prior to completing two cycles of treatment. Phase 2 will evaluate anti-tumor activity and safety of the RP2D determined during Phase 1b. Phase 2 will focus on a specific tumor type identified during Phase 1/1b and will enroll approximately 30 patients.

Safety will be monitored by the Safety Review Committee (SRC) at each dose escalation in Phase 1 and at regular intervals throughout Phase 1b and Phase 2.

Overall Response Rate (ORR), Progression Free Survival (PFS), Response Rate (RR), Overall Survival (OS), Disease Control Rate (DCR), and Complete and Partial response (CR and PR) will be used to evaluate efficacy per RECIST v1.1 criteria based on the results of positron emission tomography and computed tomography (PET-CT), computerized tomography (CT), and magnetic resonance imaging (MRI) scans.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written consent on an Informed Consent Form (ICF), approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific evaluation. Patients should have the ability to read and understand the ICF, ask for any clarifications from the study staff, and be able to comply with all planned study procedures.
2. 18 years of age or older at the time of informed consent.
3. Female patients must be at least 2 years postmenopausal (defined as 2 years without menses), surgically sterile (at least 6 months prior to dosing; must be documented) or practicing effective contraception (must agree to use 2 forms of contraception, 1 of which must be a barrier method) and willing to continue to use effective contraception for the duration of study participation and for 6 months after the final dose of study drug. Female patients must be nonlactating and have a negative serum pregnancy test result at screening and baseline.
4. Male patients must agree to use effective contraception (must agree to use 2 forms of contraception, 1 of which must be a barrier method) for the duration of study participation and for 6 months after the final dose of study drug.
5. Have a histologic or cytologic diagnosis of malignant solid tumor for which there are no standard of care treatment options known to confer a clinical benefit or for which the patient is ineligible or declines.

   A. For Phase 1 dose escalation: histologic or cytologic diagnosis of malignant solid tumor of any type. The Sponsor may remove specific tumor indications based on emerging, real-time study data.

   B. For Phase 1b dose expansion:

   i. Cohort A: Histologic or cytologic diagnosis of NSLC (adenocarcinoma and SCC).

   ii. Cohort B: Histologic or cytologic diagnosis of TNBC or HR positive, HER2 negative breast cancer.

   iii. Cohort C: Histologic or cytologic diagnosis of the following advanced metastatic solid tumors refractory to standard treatment: pancreatic adenocarcinoma, gastric adenocarcinoma, hepatocellular carcinoma, ovarian adenocarcinoma, and squamous cell carcinoma including, but not limited to, primary malignancies of the head and neck, esophagus, cervix, and skin. The Sponsor may add or remove specific tumor indications based on emerging, real-time study results.
6. Availability of a tumor tissue sample (formalin-fixed paraffin embedded [FFPE]) must be confirmed for analysis of EphA5 expression based on IHC. Tumor biopsies are not required and should not be performed to assess eligibility.

   A. For Dose Escalation (Phase 1) and Dose Expansion (Phase 1b), tumor EphA5 expression will not be required for enrollment.
7. For Dose Escalation (Phase 1), patients may have evaluable disease or measurable disease according to RECIST v1.1). For Dose Expansion (Phase 1b) and Phase 2, patients must have measurable disease according to RECIST v1.1.
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
9. Life expectancy ≥ 3 months as assessed by the investigator.
10. Hematologic function, as follows (no red blood cell [RBC] or platelet transfusions are allowed within 14 days of the first dose of MBRC-101):

    A. Absolute neutrophil count (ANC) ≥ 1.0 × 109/L B. Platelet count ≥ 100 × 109/L C. Hemoglobin ≥ 9 g/dL
11. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min by the CKD-EPI or similar equation or as measured by 24-hour urine collection.
12. Total bilirubin ≤ 1.5 × upper limit normal (ULN).
13. AST ≤ 3.0 × ULN.
14. ALT ≤ 3.0 × ULN.
15. International normalised ratio (INR) < 1.5 (or ≤ 3.0 if on therapeutic anticoagulation).
16. Treatment with other agents for cancer, if received, must have been discontinued ≥ 2 weeks prior to first dose of study drug.

Prior ADC therapy is allowed. Prior agents conjugated to MMAE are allowed for Phase 1 but not for Phase 1b or Phase 2. These exclusionary agents include brentuximab vedotin, polatuzumab vedotin, enfortumab vedotin, disitamab vedotin, tisotumab vedotin, and any MMAE-conjugated agents approved subsequent to the publication of this Protocol.

Exclusion Criteria:

1. Preexisting sensory neuropathy Grade ≥ 2.
2. Preexisting motor neuropathy Grade ≥ 2.
3. Uncontrolled central nervous system metastases.
4. Use of any investigational drug within 14 days prior to the first dose of study drug.
5. Any anticancer therapy within 14 days prior to the first dose of study drug, including: small molecules, immunotherapy, chemotherapy, monoclonal antibody therapy, radiotherapy, or any other agents to treat cancer (anti-hormonal therapy given for advanced prostate cancer or as adjuvant therapy for early stage, hormone receptor (HR) positive breast cancer is not considered cancer therapy for the purpose of this Protocol).
6. Strong CYP3A or inducers within 14 days prior to the first dose of study drug.

8. 7. Thromboembolic events and/or bleeding disorders 14 days (e.g., venous thromboembolism [VTE] or pulmonary embolism [or PE]) prior to the first dose of study drug.

8. Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class 3-4 within 6 months prior to the first dose of MBRC-101.

9. A baseline QT (time from the beginning of the Q wave to the end of the T wave) interval as corrected by Fridericia's formula (QTcF) > 470 msec.

10. Human immunodeficiency virus (HIV) infection with 1 or more of the following: A. Acquired immunodeficiency syndrome (AIDs)-defining opportunistic infection within 6 months of the start of screening; B. A change in antiretroviral therapy within 3 months of the start of screening and viral load > 500 copies/mL; C. Receiving antiretroviral therapy that may interfere with study drug; D. CD4 count < 350 at screening. 11. Active or symptomatic viral hepatitis. Patients who have been properly treated for hepatitis C infection can be included if they do not have active hepatitis C.

12. Known sensitivity to any of the ingredients of the investigational product MBRC-101.

13. Major surgery within 28 days prior to first dose of study drug. 14. History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Allowed exceptions are patients with: A. Non-melanoma skin cancer considered completely cured; B. Localized prostate cancer treated with curative intent with no evidence of progression; C. Low-risk or very low-risk (per standard clinical guidelines) localized prostate cancer under active surveillance without immediate intent to treat; D. Malignancy that is otherwise considered cured with minimal risk of recurrence.

15. Currently receiving systemic antimicrobial treatment for active infection (bacterial, viral, or fungal) at the time of first dose of MBRC-101. Routine antimicrobial prophylaxis is permitted.

16. Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study.

17. Any medical, psychiatric, addictive, or other kind of disorder which compromises the ability of the patient to give written informed consent and/or to comply with procedures.

18. Active ocular surface disease at baseline or any components of the ophthalmologic history which, in the investigator's opinion, may place the patient at significant risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse events (TEAEs) | Up to 24 Months
  TEAEs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.5.0.
Occurrence of dose limiting toxicities (DLTs) during the DLT evaluation period | 21 Days
  The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 Months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to the response evaluation criteria in solid tumors (RECIST) version 1.1.
Duration of Response (DOR) | Up to 24 Months
  DOR will be calculated among responders (PR or better) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease per RECIST version 1.1 response criteria, or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) | Up to 24 Months
  PFS will be calculated from the date of first dose of MBRC-101 to the date of first documented evidence of progressive disease as defined by RECIST version 1.1 response criteria or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 24 Months
  DCR will be defined as the proportion of patients with best overall response of Complete Response, Partial Response, or Stable Disease (SD) according to the response evaluation criteria in solid tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado, Anschutz Cancer Pavilion (ACP(, Aurora, Colorado
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Horizon Oncology Research, Lafayette, Indiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - PRISMA Health, Institute for Translational Oncology, Greenville, South Carolina
  - NEXT Oncology, Austin, Texas
  - NEXT Oncology, Irving, Texas
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staquicini FI, Tang FH, de Oliveira V, Kim SY, Chen ER, Markosian C, Staquicini DI, Wu Y, Parsons JK, Barnhart KF, Alley SC, Chen I, Arap W, Pasqualini R. First-generation and preclinical evaluation of an EphA5-targeted antibody-drug conjugate in solid tumors. J Clin Invest. 2025 Jul 15;135(14):e188492. doi: 10.1172/JCI188492. eCollection 2025 Jul 15. PMID 40662373